CLINICAL TRIAL: NCT04984291
Title: Zimmer Biomet Shoulder Arthroplasty Long-term Post Market Clinical Follow-up Study
Brief Title: Zimmer Biomet Shoulder Arthroplasty PMCF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMU2019-35E
Record Dates: First submitted 2021-07-16; First posted 2021-07-30 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Shoulder Fractures; Shoulder Arthritis; Shoulder Osteoarthritis; Shoulder Deformity; Shoulder Injuries; Shoulder Pain
Keywords: Total Shoulder Arthroplasty; Glenoid; Humeral Stem; Stem Adapter; Humeral Head; Humeral Bearing; Humeral Trays; Head Adapter; Reverse; Anatomic; Hemi
MeSH Terms: conditions — Shoulder Fractures; Shoulder Injuries; Shoulder Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Zimmer Biomet Total Shoulder Arthroplasty System (Experimental): Patients who are having primary or revision total shoulder arthroplasty who will receive a Zimmer Biomet Total Shoulder Arthroplasty System.
  Interventions: Device: Alliance Glenoid; Device: Identity Stem

INTERVENTIONS:
Device: Alliance Glenoid — Alliance Glenoid used in Primary or Revision Total Shoulder Arthroplasty
  Other Names: Alliance
Device: Identity Stem — Identity Shoulder System is intended to be used in anatomic total shoulder arthroplasty, shoulder hemi-arthroplasty, or total reverse shoulder arthroplasty in both Primary or Revision Total Shoulder Arthroplasty
  Other Names: Identity

SUMMARY:
The objectives of this study are to confirm the safety, performance, and clinical benefits of Zimmer Biomet Shoulder Arthroplasty Systems and its instrumentation in primary or revision shoulder arthroplasty. These objectives will be assessed using standard scoring systems, radiographic evidence, and adverse event records. Safety of the system will be assessed by monitoring the frequency an incidence of adverse events.

DETAILED DESCRIPTION:
The primary endpoint is defined as survival of the implant at 10 years, which is based on removal or intended removal of at least 1-study implant component and will be determined by using the Kaplan Meier method. The safety of the system will be assessed by monitoring the frequency and incidence of adverse events. Separate analysis will be done for each arm of the study.

The secondary endpoint is represented by the performance and clinical benefits of Zimmer Biomet Shoulder Arthroplasty Systems and its instrumentation after 2 years, which will be assessed by the American Shoulder and Elbow Surgeons (ASES) shoulder score. The secondary endpoint evaluation will also assess the overall pain, functional performance, quality of life and radiographic parameters of all enrolled study subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 20 years of age or older.
* Patient must be anatomically and structurally suited to receive shoulder arthroplasty implants.
* Patient is a candidate for shoulder arthroplasty due to one or more of the following:

  * Non-inflammatory degenerative joint disease including osteoarthritis and avascular necrosis.
  * Rheumatoid arthritis.
  * Correction of functional deformity.
  * Fractures of the proximal humerus, where other methods of treatment are deemed inadequate.
  * Difficult clinical management problems, where other methods of treatment may not be suitable or may be inadequate.
* Patient must be able and willing to complete the protocol required follow-up.
* Patient must be able and willing to sign the IRB/EC approved informed consent.
* Patient has grossly deficient rotator, (for reverse application)

  * With severe arthropathy and/or
  * Previously failed shoulder joint replacement
* Patient must have functional deltoid muscle (for reverse application)

Exclusion Criteria:

* Patient is unwilling or unable to give consent or to comply with the follow-up program.
* Patient has any condition which would in the judgement of the Investigator, place the patient at undue risk or interfere with the study.
* Patient is known to be pregnant or breastfeeding.
* Patient is a vulnerable subject (prisoner, mentally incompetent or unable to understand what participation to the study entails, a known alcohol or drug abuser, and/or anticipated to be non-compliant).
* Patient is uncooperative or patient with neurologic disorders who is incapable or unwilling to follow directions.
* Patient has any sign of infection affecting the shoulder joint or in its proximity which may spread to the implant site.
* Patient has rapid joint destruction, marked bone loss, or bone resorption apparent on roentgenogram.
* Patient has any neuromuscular disease compromising the affected limb that would render the procedure unjustifiable.
* Patient presents with osteoporosis, which in the opinion of the Investigator, may limit the subject's ability to support total shoulder arthroplasty using the study device.
* Patient has osteomalacia.
* Patient has a metabolic disorder that may impair bone formation.
* Patient has deficient rotator cuff.
* Patient presents with significant injury to the upper brachial plexus.
* Patient has paralysis of the axillary nerve.
* Patient has non-functional deltoid or external rotator muscles.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Estimated)
Dates: Start 2021-07-28 (Actual); Primary Completion 2033-08-15 (Estimated); Study Completion 2033-08-15 (Estimated)

PRIMARY OUTCOMES:
Implant Survivorship at 10 years follow-up (Kaplan Meier) | 10 years
  Based on removal or intended removal of the device and determined using the Kaplan-Meier method.
Frequency and Incidence of Adverse Events (Safety) | 10 years
  Monitoring the frequency and incidence of adverse events, serious adverse events, adverse device effects, serious adverse device effects, and unanticipated serious adverse device effects as well as device deficiencies.

SECONDARY OUTCOMES:
Clinical efficacy of the device is assessed using the American Shoulder and Elbow Surgeons (ASES) Shoulder Score at 2 years follow-up | 2 years
  Pain, function, and activities of daily living are measured. The ASES scale is 0-100. 100 is the highest score and indicates the greatest function while 0 is the lowest score.
Euroqol Patient Quality of life measured at 2 years follow-up (EQ-5D-5L) | 2 years
  The EuroQol five dimensions questionnaire (EQ-5D-5L) is a five dimensional self-assessment that is comprised of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. These five dimensions can be used to index a subject's health utility on a scale of 0 to 1, where 0 is death and 1 is perfect health. The scoring rule for EQ-5D permits scores less than 0, implying that some health states may be worse than death.
Radiographic Performance [Radiolucency] at 2 years follow-up | 2 years
  X-rays will be evaluated for radiolucency lines to show the number of subjects with radiolucency. Radiolucency refers to structures that are less dense and permit the x-ray beam to pass through them. Radiolucent structures appear dark or black in the radiographic image.
Radiographic Performance [Osteolysis] at 2 years follow-up | 2 years
  X-rays will be evaluated for osteolysis to show the number of subjects with osteolysis. Osteolysis is a progressive condition where bone tissue is destroyed. In this process, bones lose minerals (mostly calcium), softens, degenerates and become weaker.
Radiographic Performance [Heterotopic Ossification] at 2 years follow-up | 2 years
  X-rays will be evaluated for heterotopic ossification to show the number of subjects with heterotopic ossification. Heterotopic ossification refers to the presence of bone in soft tissue where bone normally does not exist (extraskeletal bone).
Radiographic Performance [Humeral Component Subsidence] at 2 years follow-up | 2 year
  X-rays will be evaluated for humeral component subsidence to show the number of subjects with subsidence. Component Subsidence refers to the presence of the device component gradually sinking or caving into the bone structure.
Radiographic Performance [Glenoid Component Migration] at 2 years follow-up | 2 year
  X-rays will be evaluated for glenoid component migration to show the number of subjects with migration. Component migration refers to the presence of the device component gradually moving anteriorly, posteriorly, superiorly, or inferiorly in relation to original placement.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Boylan, Study Director — Zimmer Biomet
Locations (17):
- United States (12):
  - Hoag Orthopedic Institute, Irvine, California
  - Panorama Orthopaedic and Spine Center, Golden, Colorado
  - Northwestern University, Chicago, Illinois
  - Norton Healthcare, Inc, Louisville, Kentucky
  - William Beaumont Hospital, Royal Oak, Michigan
  - TRIA Orthopaedic Center Research Institute, Bloomington, Minnesota
  - Mississippi Sports Medicine and Orthopaedic Center, PLLC, Jackson, Mississippi
  - Advance Bone and Joint, City of Saint Peters, Missouri
  - Washington University, St Louis, Missouri
  - University of Buffalo, Buffalo, New York
  - Rothman Institute, Philadelphia, Pennsylvania
  - Intermountain Health, Murray, Utah
- Japan (4):
  - Fukui General Hospital, Fukui
  - Iwaki City Medical Center, Fukushima
  - Yuuai Medical Center, Okinawa
  - Kichijoji Minami Hospital, Tokyo
- Kensington Private Hospital, Whangarei, New Zealand